CLINICAL TRIAL: NCT05591885
Title: The Effect of Nutrilite Memory Builder on the Improvement of Cognitive Function: A Randomized Controlled Trial(RCT)
Brief Title: Nutrilite Memory Builder on the Improvement of Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IS20220006RD
Record Dates: First submitted 2022-10-12; First posted 2022-10-24 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Function
Keywords: MMSE; MoCA; WMS-R; Cognitrax Test

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial:The study center will recruit 100 male or female subjects aged 40-75 years as needed. Enrolled subjects will be divided into 2 groups, with 50 subjects in each group. Study subjects will be administrated with either the Amway product or a placebo for three months (12 weeks). At least 42 subjects in each group (84 in total) are required to complete the study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study product gruop (Experimental): Nutrilite Memory Builder Ingredients (Cistanche deserticola extract, Ginkgo biloba extract, glucose, microcrystalline cellulose, corn starch, etc.) 60 Tablets / bottle
  Interventions: Dietary Supplement: Study product group (Nutrilite Memory Builder)
- Placebo group (Placebo Comparator): Ingredients (glucose, microcrystalline cellulose, corn starch, caramel pigment, etc.) 60 Tablets / bottle
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Study product group (Nutrilite Memory Builder) — During study intervention, subjects are required to take the randomly assigned study product following the instructions.Take one tablet twice daily with meals.
  Arms: Study product gruop
Dietary Supplement: Placebo group — During study intervention, subjects are required to take the randomly assigned placebo following the instructions.Take one tablet twice daily with meals.
  Arms: Placebo group

SUMMARY:
Its a randomized controlled trial, to evaluate the effect of NUTRILITE Memory Builder on the improvement of cognitive function in middle-aged and elderly people.

DETAILED DESCRIPTION:
The study center will recruit 100 male or female subjects aged 40-75 years as needed. Enrolled subjects will be divided into 2 groups, with 50 subjects in each group.

Study subjects will be administrated with either the Amway product or a placebo for three months (12 weeks). At least 42 subjects in each group (84 in total) are required to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 40-75 years old (with age groups of 40-60 years and 61-75 years as close as possible to a 1:1 ratio);
* Healthy subjects with no underlying diseases and no drug treatment at the time of screening;
* Meet the requirements of MMSE scores of 24-29;
* Be willing to comply with all study requirements and procedures;
* Agree to sign the informed consent form.

Exclusion Criteria:

* Participated in similar clinical trials in the last 6 months;
* Have mental illness or disorders of consciousness and behavior;
* Have severe chronic diseases and are currently under treatment with drugs;
* Have taken drugs that can affect cognitive function (such as first-generation antihistamines, benzodiazepines, sedatives, opiates, stabilizers, antidepressants, cholinergic drugs, anticholinergic drugs, prescription anti-inflammatory drugs) and any other regularly influential agents.
* Had flu/virus symptoms within 3 months before screening;
* Received within 3 months before screening or currently receiving medical or nutritional treatments, including protein supplementation or substances that provide exercise capacity;
* Had weight gain or weight loss of more than 5kg within 3 months before screening;
* Have a history of hospitalization within 3 months before screening;
* Have any of the following medical history or have been clinically diagnosed with any of the following diseases: obvious gastrointestinal disorders; liver, kidney, endocrine, blood, respiratory and cardiovascular diseases. These may affect the assessment of product efficacies.
* Have high daily alcohol consumption, i.e. more than 14 bottles of beer (350 ml/bottle) or wine (180 ml/bottle) per week;
* The PI believes that the subjects cannot fully cooperate with the trial arrangement.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | endpoint( day 90)
  Change of mental status after 90-days product intervention
Wechsler Memory Scale RC | endpoint( day 90)
  Change of memory after 90-days product intervention. A complete set of memory evaluation tools with 10 subscales measured three aspects of participants' long-term, short-term and instantaneous memory, which added three sub-tests to WMS. Among them, there are 3 sub-tests of long-term memory, namely personal experience, orientation, and numerical order; There are 6 sub-tests for short-term memory, namely visual rerecognition, picture recall, visual regeneration, associative learning, touch, and comprehension; Instantaneous memory has only 1 sub-test, i.e. reciting numbers in a forward and backward manner. Scoring uses the Memory Quotient (MQ) method, where higher MQ values indicate better memory ability.

SECONDARY OUTCOMES:
Quality of Life Scale | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Record the data of the subjects' life quality,The quality score is 60 points, the good is 51-60 points, the good is 41-50 points, the general is 31-40 points, the poor is 21-30 points, and the quality of life is < 20 points.
Activities of Daily Living Scale | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Record the data of the subjects' activities of daily living；The scoring results can be divided into four grades: grade 0=self-care: 100 points, good ability of daily living activities, without help from others grade=mild dysfunction: 99-61 points, able to independently complete some daily activities, but need help; Level II=moderate dysfunction: 60-41 points, need great help to complete activities of daily living Level III=severe dysfunction: ≤ 40 points, most activities of daily living can not be completed completely need care.
Verbal Memory Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' verbal memory
Finger Tapping Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' finger movement
Symbol Digit Coding Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' processing speed, working memory, visuospatial processing, and attention.
Stroop Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' memory and attention.
Shifting Attention Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' measures the subject s ability to shift from one instruction set to another quickly and accurately.
Continuous Performance Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' different aspects of attention.
Four-part Continuous Performance Test of Cognitrax Test | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Use the official website(www.cnsvs.com) to test subjects' cognitive ability.
Montreal Cognitive Assessment; | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Test Cognitive Ability
72-hrs Food Recall | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  72-hours food recall of subjects
Sport Frequency Questionnaire | baseline(day 0)/interim ( day 45)/endpoint( day 90)
  Record the exercise frequency and duration within one week, without any score.
Blood | baseline(day 0)/endpoint( day 90)
  blood routine test （red blood cell count, white blood cell count, platelet count，hemoglobin）
Urine | baseline(day 0)/endpoint( day 90)
  Urine routine test（Leukocyte, Urine Protein, Ketone Body）

CONTACTS AND LOCATIONS:
Overall Officials: Wenan Wang, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Kangrong Clinic, Jinhua, Zhejiang, China